CLINICAL TRIAL: NCT05182346
Title: Acupressure of Acupoints Versus Ischemic Compression Release of Myofascial Trigger Points in Non-specific Neck Pain: Randomised Controlled Trial
Brief Title: Acupressure Versus Ischemic Release in Non-specific Neck Pain
Acronym: Manual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soheir Shehata RezkAllah Samaan (Other)
Responsible Party: Sponsor-Investigator, Soheir Shehata RezkAllah Samaan, Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CURs; Reaserch promotion (Other: Faculty of Physical Therapy)
Record Dates: First submitted 2021-11-10; First posted 2022-01-10 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Manual Therapy; Neck Pain
Keywords: Acupressure; Ischemic Compression Release; Neck Pain.
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupressure of classical acupoints (Experimental): Acupressure is applied on four acupoints: Pressure was applied to large intestine 10 (LI10) (large intestine meridians): It is located on the dorsal radial side of the forearm, 2 Cun below the transverse cubital crease. Hegu (large intestine meridians, LI 4): It is in the middle of the 2nd metacarpal bone on the radial side. TE5 (Triple energizer): It is located 2 cun proximal to the dorsal wrist crease between the radius and the ulna. SI3 (small intestine meridians): It is located at the ulnar end of the distal palmar crease proximal to the 5th metacarpal phalangeal joint. These acupoints are commonly used in the treatment of cervical myofascial pain syndrome.
  Interventions: Procedure: Manual therapy
- Ischemic compression release of myofascial trigger points (Experimental): Ischemic compression was gradually applied pressure to the trigger point with your thumb. The patient will likely feel referred pain in a question mark pattern (along the back of the neck, around the side of the head, and then a focused pain right behind the eye). Keep in communication with the patient, checking to ensure that in staying within the limits of his pain tolerance. Hold this technique for approximately 20 seconds to 1 minute, patient tells you that pain has diminished, or until feels the muscle fibers begin to relax under your pressure. Once feel this release, gradually release pressure. All identified trigger points will be treated. Then apply a few effleurage strokes to flush out the area and follow up with a passive stretch to the muscle.
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Procedure: Manual therapy — * Acupressure of acupoints is manipulation of classic acupoints by pressure.
  * Ischemic compression release is applying pressure to the myofascial trigger points until release of these points.
  Other Names: Acupressure; Ischemic compression release

SUMMARY:
Chronic neck pain (CNP) attributed to myofascial pain syndrome (MFPS) which is one of the particularly common skeletal muscle disorder associated with the hyperirritable zone in the taut band of muscle. Myofascial trigger points (MTrP) are one of the most overlooked and ignored causes of musculoskeletal pain. This study aims to compare the clinical efficacy of acupressure of cervical acupoints versus ischemic compression release (ICR) of MTrPs in CNP.

DETAILED DESCRIPTION:
Nonspecific neck pain (NSNP) is the commonest cause of neck symptoms and results from postural and mechanical causes.Chronic neck pain (CNP) attributed to myofascial pain syndrome (MFPS) which is one of the particularly common skeletal muscle disorder associated with the hyperirritable zone in the taut band of muscle. Myofascial trigger points (MTrP) are one of the most overlooked and ignored causes of musculoskeletal pain.The objectives of this study is to compare the clinical efficacy of acupressure of cervical acupoints versus ischemic compression release (ICR) of MTrPs in CNP. This single blind randomized trial involves patients with NSNP were randomly assigned into three groups: the acupressure group (ACG), and the ischemic compression release group (ICRG) and the control group (CG). Patients in all groups received hot packs and post-isometric relaxation. Patients in ACG received acupressure at local acupuncture points, Gall bladder 21 (GB 21), small intestine 14 (SI 14) and SI 15, and the ICRG received pressure on MTrPs of trapezius muscle on both sides. VAS sores, pressure pain threshold (PPT), neck lateral flexion range of motion, and neck disability index (NDI) were assessed before and after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All participants have nonspecific NP for a period of >3 months
* All participants are presented with at least one active MTrP at the upper trapezius muscle, -
* All participants had not used any medications or physiotherapy to alleviate pain were included in this study.

Exclusion Criteria:

* Participants who met these criteria had been excluded:

  1. NP due to trauma, whiplash, cervical disc prolapse, inflammation, malignant disease, or any other neurological and orthopedic conditions, which will affect the assessment.
  2. Congenital malformation of the spine as it will alter the normal pattern of movements.
  3. Had any invasive therapies in the past month.
  4. Patients with sensory impairments, such as diabetic sensory neuropathy.
  5. Mental disorders.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-06-13 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 successive weeks
  - The Visual Analog Scale (VAS) assessed the intensity of general pain and pain in the right and left upper trapezius. The scale consists of an unanchored horizontal line 10 centimeters in length, with one end corresponding to zero ("no pain") and the other to 10 ("maximum pain").
Pressure pain threshold | 4 successive weeks
  The palpated trigger points are marked with a skin marker. The patient is positioned accordingly and a dial type pressure algometer is placed on the site and a con¬stant vertical pressure was applied to the site. The subject is instructed to express pain by raising their hands when only slight pain was felt, until then the pressure is increased at a constant rate.
Cervical range of motion | 4 successive weeks
  It was aligned on the Nose Bridge and ears and was fastened to the head by a Velcro strap. It was imperative that the patient's chair be positioned such that the magnetic field would zero the dial meter for the rotation component. Prior to testing, Subjects were instructed to sit erect in the chair, with their low back against the chair, midback away from the chair, arms hanging at sides, and feet flat on the floor. Active right and left lateral flexion components of cervical spine motion were measured twice on each subject. During testing, all dials read zero before the desired component was measured. A horizontal line was placed on the wall for the purpose of tracking; subjects were instructed to follow this line when the lateral flexion component was measured

SECONDARY OUTCOMES:
Neck function | 4 successive weeks
  The neck disability index is composed of ten descriptions which assess an individual's daily activities, pain and concentration in regards to their functional sta¬tus. Each question carries six responses on a scale of 0-5 (Howard, 1991). The maximum possible score is 50. Disability is cal¬culated using the NDI raw score as no disability (0-4), mild (5-14), moderate (15-24), severe (25-34) and complete (<34).The Neck Disability Index (NDI) is the most widely used instrument in neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Soheir S RezkAllah, professor, Study Chair — Professor of physical therapy, Cairo University
Locations (1):
- Soheir, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim M, Kim J. Effects of Acupressure on Pain, Flexibility, and Substance P in Middle-Age Women with Chronic Neck Pain. J Altern Complement Med. 2021 Feb;27(2):160-167. doi: 10.1089/acm.2020.0413. Epub 2020 Dec 8. PMID 33296258